CLINICAL TRIAL: NCT07212205
Title: The Effect of Visual and Auditory Cueing Walker on Gait in Individuals With Parkinson's Disease Experiencing Freezing of Gait
Brief Title: Freezing in Parkinson's Disease
Acronym: parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Asst. Prof., Necmettin Erbakan University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: nezahat keleşoğlu; Necmettin Erbakan university (Other: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Auditory and Visual cue; Gait; Parkinson's disease; Walker
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Arm 1: PDF (Parkinson's Disease with Freezing of Gait)
  Intervention: Visual & Auditory Cueing Walker
  Description: Participants were assessed under two within-subject conditions: walking without cues and walking with a visual & auditory cueing walker.
  Arm 2: PDNF (Parkinson's Disease without Freezing of Gait)
  Intervention: Visual & Auditory Cueing Walker
  Description: Participants were assessed under two within-subject conditions: walking without cues and walking with a visual & auditory cueing walker.
  This is a non-randomized interventional study with two parallel groups (PDF and PDNF). Each participant was assessed under two within-subject conditions: walking without cues and walking with a visual and auditory cueing walker. The two conditions are repeated measures within each arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDF (Parkinson's Disease with Freezing of Gait) (Experimental): Intervention Name: Visual & Auditory Cueing Walker
  Description:
  "Participants in this arm were assessed under two within-subject conditions: walking on a 7-meter path without cues (control condition) and walking on the same path using a visual and auditory cueing walker (intervention condition). Each participant completed both conditions in a single session. Pre- and post-walking evaluations were conducted for walking speed (Timed Up and Go Test), fall risk (Tinetti Balance and Gait Assessment), and gait adaptation (Dynamic Gait Index). The 'no cues' condition represents a repeated-measures control within the same arm. Participants were included based on the presence of freezing of gait."
  Planned Enrollment: 18
  Interventions: Other: Visual & Auditory Cueing Walker
- PDNF (Parkinson's Disease without Freezing of Gait) (Experimental): Intervention Name: Visual & Auditory Cueing Walker
  Description:
  "Participants in this arm were assessed under two within-subject conditions: walking on a 7-meter path without cues (control condition) and walking on the same path using a visual and auditory cueing walker (intervention condition). Each participant completed both conditions in a single session. Pre- and post-walking evaluations were conducted for walking speed (Timed Up and Go Test), fall risk (Tinetti Balance and Gait Assessment), and gait adaptation (Dynamic Gait Index). The 'no cues' condition represents a repeated-measures control within the same arm. Participants were included based on the absence of freezing of gait."
  Planned Enrollment: 12
  Interventions: Other: Visual & Auditory Cueing Walker

INTERVENTIONS:
Other: Visual & Auditory Cueing Walker — Intervention Name:
  Visual & Auditory Cueing Walker
  Other Intervention Names (varsa):
  Cueing Walker Walker with Visual & Auditory Cues
  Intervention Description:
  "Participants in this arm were assessed under two within-subject conditions: walking on a 7-meter path without cues (control condition) and walking on the same path using a visual and auditory cueing walker (intervention condition). Each participant completed both conditions in a single session. Pre- and post-walking evaluations were conducted for walking speed (Timed Up and Go Test), fall risk (Tinetti Balance and Gait Assessment), and gait adaptation (Dynamic Gait Index). The 'no cues' condition represents a repeated-measures control within the same arm. Participants were included based on the presence of freezing of gait."
  Planned Enrollment: 18

SUMMARY:
The aim of this study was to investigate the effects of a visual and auditory cueing walker on freezing of gait during walking in patients with Parkinson's disease (PDF), compared to Parkinson patients without freezing of gait (PDNF).Sample size was calculated to detect a difference of 0.37 m/sec on mean velocity, with a deviation of 0.3 m/sec, two-sided 5% significance level, and power of 90%. Considering the expected 10% dropout rate, twelve subjects were included.Researcher R1 determined whether the subject was eligible for inclusion in the trial and researcher R2 carried out the gait analysis. Both examiners were unaware of group allocation. An independent researcher (R3) performed the clinical evaluation before the procedures started. Participants walked back and forth on a 7-meter walking path under two different conditions: without cues and with a walker providing visual and auditory cues. To assess the risk of falls in both groups, the "Tinetti Balance and Gait Assessment" was conducted. Additionally, the "Dynamic Gait Index" was used to evaluate the ability to adapt walking to varying task demands, and the Timed Up and Go Test (TUGT) was employed to determine walking speed.

DETAILED DESCRIPTION:
This study suggests that a walker providing visual and auditory cues may improve daily walking in patients with Parkinson's disease with freezing of gait (PDF) and reduce the risk of falls in patients with Parkinson's disease without freezing of gait (PDNF) who exhibit hypokinetic gait patterns.

ELIGIBILITY:
Inclusion Criteria:Those with a Hoehn-Yahr classification between 2.5 and 4 were included in the study.

-

Exclusion Criteria:Patients with secondary parkinsonism, severe systemic diseases, psychiatric illness, cognitive impairment (Mini-Mental State Examination score <24), hearing and vision loss, musculoskeletal problems, or symptoms suggestive of cerebellar dysfunction were excluded from the study.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Gait Adaptation | Immediately after walking with the visual and auditory cueing walker test was completed
  Dynamic Gait Index: Time taken by the participant to complete the 7-meter walking path under each condition (without cues and with visual & auditory cueing walker), measured using the Timed Up and Go Test (TUGT).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Meram
  - Necmettin Erbakan University, Konya, Meram

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to participant privacy and confidentiality concerns, as well as institutional regulations governing sensitive patient information.